CLINICAL TRIAL: NCT04463069
Title: School-based Physical Activity Intervention for Obesity Among Adolescents With Intellectual Disability in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Gao Yang, Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30160054
Record Dates: First submitted 2020-06-28; First posted 2020-07-09 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Obesity
Keywords: adolescents; intellectual disability; overweight; obesity; physical activity; intervention
MeSH Terms: conditions — Obesity; Intellectual Disability; Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in the intervention group participated in the APA intervention consisting of simple and fun endurance and strength-building exercise at a frequency of two sessions per week.
  Interventions: Other: Adapted physical activity
- control group (No Intervention): Participants in the control group received no intervention in the study time period.

INTERVENTIONS:
Other: Adapted physical activity — This PA program was modified from an adapted physical activity (APA) program that designed for obesity management among adolescents with intellectual disability (ID). The aim of the APA program was to promote PA and health for people in special needs. In this study, the APA program was carefully designed based on a comprehensive pre-intervention assessment of each adolescent with ID, so that can be able to address their individual needs in learning and adaption. The APA program comprised three stages of APA training at school and each stage consisted of simple and fun endurance and strength-building exercise, at a frequency of two sessions per week, and lasting for about three months.
  Arms: intervention group

SUMMARY:
Considering that children with intellectual disability (ID) might be more vulnerable to obesity than their counterparts in the general population. This study aimed to develop and evaluate the effectiveness of an adapted physical activity (APA) program in reducing weight among adolescents with ID. The hypothesis of the study was the APA program would be able to decrease obesity among adolescents with ID.

DETAILED DESCRIPTION:
Background: Children with intellectual disability (ID) might be more vulnerable to obesity than their counterparts in the general population. This study aimed to evaluate the effectiveness of an adapted physical activity (APA) program in reducing weight among adolescents with ID.

Methods: A 9-month randomized controlled trial of a school-based APA program was conducted in adolescents with ID and overweight/obesity in Hong Kong. The intervention group received the APA program which consisted of endurance and strength-building exercises at a frequency of two sessions per week, while the control group received routine PE classes as usual. Data on obesity-related variables were collected before the intervention, at the midpoint of the intervention and after the intervention. Linear mixed-effect models were used to examine the intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* aged between 12 and 18 years
* overweight and obesity
* mild or moderate intellectual disability

Exclusion Criteria:

* physical disability
* medical predispositions towards obesity (genetic syndrome or drug treatment)
* contraindications (e.g. asthma, heart disease)
* having participated in other exercise programs in the past 6 months.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Gao, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Hong Kong Bapist University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially, 81 eligible students with parental informed consent were recruited (41 in intervention and 40 in control). 13 in control withdrew after learning the assignment results. 5 more were then recruited into the control to fulfill sample size (32). After commencement of study, 2 and 10 withdrew from intervention and control respectively. Finally, 61 (39 in intervention and 22 in control) completed the study.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 41 | 45
Completed | 39 | 22
Not Completed | 2 | 23
Not completed — Withdrawal by Subject | 2 | 10
Not completed — Participants' parents refused to participate after learning the assignment results | 0 | 13

BASELINE CHARACTERISTICS:
Population: The analysis was performed on subjects who completed the entire study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 39 | 22 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 22 | 61
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 31 | 14 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 39 | 22 | 61

OUTCOME MEASURES:

1. Primary Outcome: BMI Change
Description: The primary outcome variable was change in BMI (weight (kg) / height2 (m)) that was further calculated from the height and weight measured at school in the morning time. Height was measured to the nearest 0.1 cm using a stadiometer and weight was measured to the nearest 0.1 kg on a TANITA digital scale (TBF-410) with the subject wearing lightweight clothing and no shoes.
Time Frame: Change from baseline at 4 months and 9 months
Measure: Mean (95% Confidence Interval); unit: kg/m2
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 22
kg/m2
  Mean change from baseline to 4 months | -0.14 [-0.44 to 0.16] | 0.42 [0.12 to 0.73]
  Mean change from baseline to 9 months | -0.66 [-1.06 to -0.25] | 0.68 [0.16 to 1.20]

2. Secondary Outcome: BMIz Change
Description: The BMIz was converted from the BMI values using WHO 2007 reference standards. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values denote a higher BMI.
Time Frame: Change from baseline at 4 months and 9 months
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 22
z-score
  Mean change from baseline to 4 | -0.06 [-0.12 to -0.00] | 0.07 [-0.00 to 0.14]
  Mean change from baseline to 9 | -0.23 [-0.32 to -0.14] | 0.10 [-0.03 to 0.22]

3. Secondary Outcome: Weight Change
Description: Weight was measured to the nearest 0.1 kg on a calibrated TANITA digital scale (TBF-410) with the subject wearing lightweight clothing and no shoes.
Time Frame: Change from baseline at 4 months and 9 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 22
kg
  Mean change from baseline to 4 | 0.42 [-0.28 to 1.12] | 1.79 [0.90 to 2.68]
  Mean change from baseline to 9 | -0.15 [-1.06 to 0.75] | 2.76 [1.45 to 4.07]

4. Secondary Outcome: Percent Body Fat Change
Description: Percent body fat was measured with the TANITA digital scale (TBF-410) using foot-to-foot bioelectrical impedance analysis.
Time Frame: Change from baseline at 4 months and 9 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 22
percent change
  Mean change from baseline to 4 | -0.19 [-1.18 to 0.80] | 0.80 [-0.24 to 1.84]
  Mean change from baseline to 9 | -1.46 [-2.41 to -0.52] | 0.24 [-0.60 to 1.07]

5. Secondary Outcome: Waist Circumference Change
Description: Waist circumference (cm) was measured with a flexible meter ribbon accurate to 0.1 cm at the midway between the lowest rib margin and the top of the iliac crest at the end of gentle expiration
Time Frame: Change from baseline at 4 months and 9 months
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 22
cm
  Mean change from baseline to 4 | -1.66 [-3.02 to -0.29] | 1.50 [-0.01 to 3.01]
  Mean change from baseline to 9 | -2.02 [-3.80 to -0.23] | 1.76 [-0.25 to 3.77]

6. Secondary Outcome: Waist-to-height Ratio Change
Description: Waist-to-height ratio was calculated by dividing the waist circumference by the height.
Time Frame: Change from baseline at 4 months and 9 months
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 39 | 22
ratio
  Mean change from baseline to 4 | -0.01 [-0.02 to -0.00] | 0.01 [-0.00 to 0.02]
  Mean change from baseline to 9 | -0.02 [-0.03 to -0.01] | 0.01 [-0.01 to 0.02]

7. Secondary Outcome: Cardiorespiratory Fitness Change
Description: Cardiorespiratory fitness was assessed using the 9-minute run/walk test. The test measured how far a person can cover a flat surface 25 meters in length over a 9-minute period.
Time Frame: Change from baseline at 4 months and 9 months
Reporting Status: Not Posted

8. Secondary Outcome: Muscular Strength and Endurance Change
Description: The muscular strength and endurance were measured by handgrip strength and sit-ups. The handgrip strength was measured using a dynamometer (Takei, TKK5001, GRIP-A digital dynamometer). The sit-ups measured the total number of correctly completed sit-ups performed in 30 seconds.
Time Frame: Change from baseline at 4 months and 9 months
Reporting Status: Not Posted

9. Secondary Outcome: Flexibility Change
Description: Flexibility was measured by the sit-and-reach test.
Time Frame: Change from baseline at 4 months and 9 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 9 months
Description: Possible adverse effects (e.g., sports injury, underweight, binge eating) suggested by previous studies will be prevented via diverse means (e.g., to inform children and parents of the possible adverse consequences in advance and provide feasible and practical preventive strategies to them). They can reach the research team via a hotline on an ad hoc basis. The adverse events will be monitored among participants who completed the baseline assessments.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/29
Other Adverse Events (participants affected / at risk) | 0/41 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT04463069/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT04463069/ICF_001.pdf